CLINICAL TRIAL: NCT06680895
Title: An Observational Study of Fractional Exhaled Nitric Oxide Concentration in Patients With Advanced Respiratory Support
Brief Title: FeNO Observation Study in ICU Patients With ARS
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiZhongshanICU
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Compare the Concentration of Exhaled Nitric Oxide in Patients With Different Severity of RF

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FeNO Observation — FeNO was observed and measured among patients with advanced respiratory support

SUMMARY:
1. Main Objective: To compare the concentration of exhaled nitric oxide in patients with different severity of respiratory failure in ICU.
2. Secondary Purpose:

   1. To observe the change of nitric oxide concentration in exhaled breath of patients with mechanical ventilation over time;
   2. The relationship and differences between pulmonary ventilation blood flow levels in patients with different exhaled NO concentrations;
   3. Reactivity of patients with different exhaled NO concentrations to inhaled nitric oxide therapy and the relationship between them.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years of age) with mechanical ventilation or advanced respiratory support in the ICU, regardless of gender;
2. The expected mechanical ventilation time of tracheal intubation is more than 24 hours;
3. The initial ventilator Settings of clinical routine were adopted: oxygen fraction (FIO2) = 50%, respiratory rate = 15/min, positive end-expiratory pressure (PEEP) = 5 cmH2O, tidal volume = 6-8 ml/kg ideal body weight (IBW), inspiration-exhalation ratio =1:2;
4. Agree to participate in this experiment and sign the informed consent.

Exclusion Criteria:

* 1.Use of any NO-containing drugs (such as nitroglycerin), anti-inflammatory drugs, or drugs or means that affect the airway diameter within 6 hours before the first FeNO measurement; 2. Participating in other clinical research projects; 3. Patients deemed unsuitable by the investigators.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU patients with advanced respiratory support
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
FeNO concentration | 1.5 year
  Exhaled nitric oxide concentration of patients with different severity of respiratory failure in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, Doctor, Study Director — Fudan University
Locations (1):
- Shanghai Zhongshan hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided